CLINICAL TRIAL: NCT00438945
Title: The Effect of Eprosartan in Patients With Essential Hypertension on Renal Tubular Function and Vasoactive Hormones During Baseline Conditions and After Activation of the Sympathetic Nervous System.
Brief Title: The Effect of Eprosartan on Hormones and Kidney Function in Patients With Essential Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Erling Bjerregaard Pedersen, Department of Medical Research, Holstebro Hospital
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: MED.RES.HOS.2006.03.HV
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — eprosartan

INTERVENTIONS:
Drug: Eprosartan

SUMMARY:
We, the investigators at Holstebro Hospital, want to test the hypothesis that eprosartan reduces the activity of the sympathetic nervous system in patients with essential hypertension - during baseline conditions and after activation of the sympathetic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years.
* Body mass index less or equal to 30 kg/m2.
* Women must use oral hormonal anticonceptive drugs, use intrauterine anticonceptive device, be sterilized / hysterectomized or be postmenopausal.
* Arterial hypertension, defined by 24 hour ambulatory blood pressure above 125 mmHg systolic or above 80 mmHg diastolic.

Exclusion Criteria:

* History of myocardial infarction.
* History of stroke.
* Heart failure.
* Endocrine organ disease.
* Lung disease.
* Clinically significant abnormal biochemical screening of the blood regarding: B-hemoglobin, P-sodium, P-potassium, P-creatinine (under 200 µmol/L will be accepted), P-albumin, p-bilirubin, p-alaninaminotransferase, P-alkaline phosphatase, p-cholesterol and B-glucose.
* Clinically significant abnormal screening of the urine regarding: albumin and glucose (protein excretion below 0.5 g/L will be accepted).
* Renovascular hypertension.
* Malignant disease.
* Alcohol abuse.
* Usage of medical drugs besides antihypertensives or statins.
* Drug abuse.
* Pregnancy or breast feeding.
* Known intolerance or allergic to eprosartan or sodium nitroprusside.
* Blood donation within 1 month of the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-01; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Heart rate
Fractional sodium excretion
Plasma levels of noradrenaline

SECONDARY OUTCOMES:
Fractional lithium excretion
Glomerular filtration rate
plasma levels of renin, angiotensin II, aldosterone, vasopressin, atrial natriuretic peptide and brain natriuretic peptide
free water clearance
urinary excretion of aquaporin 2

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, MD, professor, Study Chair — Department of Medical Research, Holstebro Hospital
Locations (1):
- Department of Medical Research, Holstebro Hospital, Holstebro, Denmark

REFERENCES:
- [Derived] Vase H, Lauridsen TG, Graffe CC, Pedersen EB. The effect of eprosartan on reflex sympathetic activation in sodium restricted patients with essential hypertension. J Am Soc Hypertens. 2011 Sep-Oct;5(5):385-94. doi: 10.1016/j.jash.2011.03.007. Epub 2011 Jun 2. PMID 21640689